CLINICAL TRIAL: NCT03048058
Title: Internet Surveys and Their Impact on Adherence and Quality of Life to Mirvaso for Rosacea
Brief Title: Internet Surveys and Their Impact on Adherence for Rosacea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00036221; NCT02659670 (obsolete NCT alias)
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Surveys and Questionnaires; Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- brimonidine topical gel 0.33% & survey (Experimental): The internet survey will ask them how often they have used their medication that week, as well as giving them treatment tips and reminders about rosacea triggers. They will be asked a variety of questions during the weekly internet survey- such as the amount of erythema they currently have (measured by VAS scale), how much burning and stinging they have, how often they have used the medication and where did they apply the medication, as well as any additional side effects they may be having from the medication.
  Interventions: Drug: brimonidine topical gel 0.33% & survey; Drug: brimonidine topical gel 0.33% & SOC
- brimonidine topical gel 0.33% & SOC (Active Comparator): Topical drug and standard of care follow-up, no weekly survey; only survey during 3 month and 6 month visits
  Interventions: Drug: brimonidine topical gel 0.33% & SOC

INTERVENTIONS:
Drug: brimonidine topical gel 0.33% & survey — The internet survey will ask them how often they have used their medication that week, as well as giving them treatment tips and reminders about rosacea triggers. They will be asked a variety of questions during the weekly internet survey- such as the amount of erythema they currently have (measured by VAS scale), how much burning and stinging they have, how often they have used the medication and where did they apply the medication, as well as any additional side effects they may be having from the medication.
  Other Names: MIRVASO
  Arms: brimonidine topical gel 0.33% & survey
Drug: brimonidine topical gel 0.33% & SOC — All subjects will receive standard-of-care brimonidine topical gel 0.33%
  Other Names: Mirvaso

SUMMARY:
An investigator-blinded, prospective, 6 month study of subjects with persistent erythema associated with active rosacea will be conducted in 20 subjects aged 18 years and older. All subjects will receive standard-of-care brimonidine topical gel, 0.33% with instructions to apply it once daily per package insert. Adherence will be assessed using weekly internet surveys to document how often the medication is being used, as well as reminders about rosacea triggers and general use of brimonidine.

DETAILED DESCRIPTION:
An investigator-blinded, prospective, 6 month study of subjects with persistent erythema associated with active rosacea will be conducted in 20 subjects aged 18 years and older. All subjects will receive standard-of-care brimonidine topical gel, 0.33% with instructions to apply it once daily per package insert. Adherence will be assessed using weekly internet surveys to document how often the medication is being used, as well as reminders about rosacea triggers and general use of brimonidine.Subjects will be randomized 1:1 to be in the weekly internet survey group or the standard care non-survey group.

At each visit, review of the internet survey use will be done to assess adherence to the medication. . Disease severity measures ((Clinician's Erythema Assessment (CEA), and Lesion counts will be obtained. QOL will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with persistent erythema associated with rosacea, age greater than 18, who agrees to participate and provide written consent.
* Have an Investigator Global Assessment of mild to moderate rosacea (IGA rating between 2 and 5 in the Investigator Global Assessment score which includes erythema in the assessment).
* Access to a computer and the internet.

Exclusion Criteria:

* Initiation or change in dose within 4 weeks of baseline of systemic anti-inflammatory medication which may influence study outcome.
* Use of topical therapy for rosacea within 2 weeks of baseline.
* Use of systemic corticosteroids within 4 weeks of baseline. Presence of a concurrent medical condition or skin condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Subjects with known allergy or sensitivity to bromonidine topical gel, 0.33% or components therein.
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile, or willing to practice effective contraception during the study. Nursing mothers, pregnant women and women planning to become pregnant while on study are to be excluded.
* Subjects with severe cardiovascular disease or vascular insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Dept of Dermatology, WFUHS, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 subjects male/female aged 18 years and older with the diagnosis of persistent erythema associated with mild to moderate rosacea as defined by an Investigator Global Assessment rating between 2 and 5. Patients were recruited from Wake Forest University Department of Dermatology Clinics and via Institutional Review Board approved advertising.
Groups:
- Brimonidine Topical Gel 0.33% & Survey: The internet survey will ask them how often they have used their medication that week, as well as giving them treatment tips and reminders about rosacea triggers. They will be asked a variety of questions during the weekly internet survey- such as the amount of erythema they currently have (measured by VAS scale), how much burning and stinging they have, how often they have used the medication and where did they apply the medication, as well as any additional side effects they may be having from the medication.
  brimonidine topical gel 0.33% & survey: The internet survey will ask them how often they have used their medication that week, as well as giving them treatment tips and reminders about rosacea triggers. They will be asked a variety of questions during the weekly internet survey- such as the amount of erythema they currently have (measured by VAS scale), how much burning and stinging they have, how often they have used the medication and where did they apply the medication,
Period: Overall Study
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Started | 10 | 10
Completed | 6 | 6
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: 20 subjects of both genders aged 18 years and older with the diagnosis of persistent erythema associated with mild to moderate rosacea as defined by an Investigator Global Assessment rating between 2 and 5.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender not collected for all participants
  Participants
    number analyzed (Participants) | 6 | 6 | 12
    Female | 6 | 6 | 12
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Adherence (% of Prescribed Doses That Were Actually Taken by the Subject)
Description: To assess adherence to topical brimonidine for the treatment of rosacea as measured by MEMS caps. The result will be the % of prescribed doses that were actually taken by the subject
Time Frame: 6 months
Measure: Median (Standard Deviation); unit: percentage of medication use
Groups:
- Brimonidine Topical Gel 0.33% & Survey: Topical drug and standard of care follow-up,with weekly survey.
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 10 | 10
percentage of medication use | 8.2 (5.3) | 6.9 (4.2)

2. Secondary Outcome: Lesion Count
Description: Change in total Lesion count
Time Frame: Baseline and 6 months
Population: Only 7 participants in the gel and survey group and 6 in the control group reported data at 6 months
Measure: Mean (Standard Deviation); unit: count of lesions
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 10 | 10
count of lesions
  Baseline | 4 (9.6) | 10.4 (17.6)
  6 Months: number analyzed (Participants) | 7 | 6
  6 Months | 2.7 (2.9) | 6.2 (6.7)

3. Secondary Outcome: Clinician Erythema Assessment Scale
Description: Clinician Erythema Assessment scale based on scale of 0-4 with 0 being no erythema and 4 being severe erythema with greater scores denoting a worse outcome.
Time Frame: baseline and 6 months
Population: Only 7 participants in the gel and survey group and 6 in the control group reported data at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 2.4 (0.5) | 2.5 (.53)
  6 Months: number analyzed (Participants) | 7 | 6
  6 Months | 2.7 (2.8) | 2.3 (.52)

4. Secondary Outcome: Quality of Life (Measured by General Survey of Impact of Rosacea on Everyday Activities)
Description: Change in overall Quality of Life as measured by the The Life Impact Survey. This measures the impact of rosacea and its treatment on life. The score range is 0-54 with higher scores denoting worse outcomes.
Time Frame: baseline and 6 months
Population: Only 7 participants in the gel and survey group and 6 in the control group reported data at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 2.4 (2.12) | 6.2 (8.66)
  6 Months: number analyzed (Participants) | 7 | 6
  6 Months | 1.43 (1.72) | 1.5 (1.05)

5. Secondary Outcome: Patient Severity Assessment (PSA)
Description: Patient Severity Assessment: Subject ratings of erythema with scale 0 - 4. 0 = face free of rosacea; 4 = My face has severe medium to large sized red inflamed bumps or pustules, My face has severe redness. Higher scores denotes worse outcomes.
Time Frame: baseline and 6 months
Population: Only 7 participants in the gel and survey group and 6 in the control group reported data at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 9 | 10
units on a scale
  Baseline | 1.6 (0.7) | 2.4 (1.26)
  6 Months: number analyzed (Participants) | 7 | 6
  6 Months | 1.14 (.9) | 1.17 (.98)

6. Secondary Outcome: Quality of Life With Rosacea
Description: Quality of life for rosacea was reported. The score range is 4-40 with higher scores denoting worse outcomes.
Time Frame: baseline and 6 months
Population: Only 7 participants in the gel and survey group and 6 in the control group reported data at 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline | 17.5 (4.25) | 13.7 (4.79)
  6 Months: number analyzed (Participants) | 7 | 6
  6 Months | 15.57 (4.35) | 13 (4.1)

7. Secondary Outcome: Dermatology Life Quality Index
Description: Dermatology Life Quality Index (DLQI) for the impact of rosacea on everyday activities. The score range is 0-30 with higher scores having a larger effect on patient's life.
Time Frame: baseline and 6 months
Population: No data was collected
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Brimonidine Topical Gel 0.33% & Survey: brimonidine topical gel 0.33% & survey adverse events
Arm/Group | Brimonidine Topical Gel 0.33% & Survey | Brimonidine Topical Gel 0.33% & SOC
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Limitations: small sample size (n=20) and poor subject retention. With limited patient data, particularly due to loss of patient follow up, the power of the study was less than ideal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03048058/Prot_SAP_000.pdf